CLINICAL TRIAL: NCT00000916
Title: A Phase II, Randomized Study of the Safety and Efficacy of Hydroxyurea in Subjects on Potent Antiretroviral Therapy With Less Than 200 Copies/ml of HIV RNA in the Plasma
Brief Title: A Study of the Safety and Effectiveness of Hydroxyurea in Patients on Potent Antiretroviral Therapy and Who Have Less Than 200 Copies/ml of HIV RNA in Their Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: A5025; 10873 (Registry Identifier: DAIDS ES); ACTG A5025
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Hydroxyurea; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; lamivudine, zidovudine drug combination; Hydroxyurea; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Hydroxyurea
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
This study compares the safety and effectiveness of continuing your current anti-HIV medications to that of adding or switching some of your anti-HIV medications. It will follow the effect of these medication changes, including the addition of hydroxyurea (HU), on long-term viral suppression. Other medications which may be added include didanosine (ddI) and/or stavudine (d4T).

Patients receiving combination antiretroviral therapy with indinavir (IDV), zidovudine (ZDV)(or d4T) and lamivudine (3TC) show viral suppression for two years or more. Discontinuation of one or two of these drugs results in prompt loss of the viral suppression. Other studies show that addition of HU to some reverse transcriptase inhibitor treatments results in increased antiviral effects. This study will provide further information on the effect of adding HU to a treatment regimen with respect to long-term viral suppression.

DETAILED DESCRIPTION:
Previous ACTG studies show that discontinuation of one or two of a three-drug regimen (IDV, ZDV, 3TC) leads to prompt loss of viral suppression in the plasma. In this trial, it will be determined whether adding hydroxyurea (HU) to a suppressive regimen increases long term viral suppression. Important safety information on the tolerance of HU regimen will be characterized in asymptomatic patients with viral suppression.

Patients are equally randomized to one of three arms and receive treatment as follows:Arm A: IDV plus ddI plus d4T plus HU placebo. Arm B: IDV plus ddI plus d4T plus HU. Arm C: IDV plus 3TC/ZDV (or d4T plus 3TC). Patients are monitored every 8 weeks with plasma HIV RNA levels and CD4 cell counts.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 13 years or older.
* Have documented HIV-1 infection.
* Are currently receiving combined IDV, ZDV(or D4T), and 3TC for at least 6 consecutive months, resulting in HIV RNA less than 200 copies/ml and CD4 cell count greater than 200 cells/mm3.
* Had a CD4 count greater than 100 cells/mm3 before starting current anti-HIV therapy.
* Are of childbearing age and agree to practice abstinence or use of combined barrier and hormonal methods of birth control during and for 3 months after the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken various medications and have various laboratory results (see technical abstract).
* Have cancer requiring chemotherapy.
* Have an unexplained fever for 7 days or diarrhea for 15 days in the month before the start of the study.
* Had prior peripheral neuropathy or hepatitis.
* Recently underwent radiation, experimental, or infection therapy.
* Are pregnant or breastfeeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 399
Dates: Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Havlir D; Richman D, Study Chair; Collier A, Study Chair; Hirsch M, Study Chair; Tebas P, Study Chair
Locations (34):
- United States (34):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Havlir DV, Gilbert PB, Bennett K, Collier AC, Hirsch MS, Tebas P, Adams EM, Wheat LJ, Goodwin D, Schnittman S, Holohan MK, Richman DD; ACTG 5025 Study Group. Effects of treatment intensification with hydroxyurea in HIV-infected patients with virologic suppression. AIDS. 2001 Jul 27;15(11):1379-88. doi: 10.1097/00002030-200107270-00007. PMID 11504959